CLINICAL TRIAL: NCT05311982
Title: Transcranial Direct Current Stimulation Modulates Spectral Power and Coherence in Autism Spectrum Disorder: a Triple-blind, Placebo-controlled Study
Brief Title: Transcranial Direct Current Stimulation in Autistic Spectrum Disorder
Acronym: TDCSinASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tdcs Autism ufpb
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Autistic Disorders Spectrum
Keywords: Autism; Tdcs; EEG
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DLPFC-L F3 (Block A) (Active Comparator): The study was developed through a triple-blind, crossover, randomized, placebo-controlled clinical trial (dummy tDCS). Participants were randomized into three groups receiving unilateral tDCS in DLPFC-L F3 (Block A)
  Interventions: Device: DLPFC-R (F4) TDCS; Device: DLPFC-L (F3) and DLPFC-R (F4) TDCS; Device: sham-tDCS
- tDCS combined in DLPFC-L (F3) and DLPFC-R (F4) (Active Comparator): The study was developed through a triple-blind, crossover, randomized, placebo-controlled clinical trial (dummy tDCS). Participants were randomized into three groups receiving unilateral tDCS in tDCS combined in DLPFC-L (F3) and DLPFC-R (F4)
  Interventions: Device: DLPFC-R (F4) TDCS; Device: DLPFC-L (F3) and DLPFC-R (F4) TDCS; Device: sham-tDCS
- Sham (Block C) (No Intervention): The study was developed through a triple-blind, crossover, randomized, placebo-controlled clinical trial (dummy tDCS). Participants were randomized into three groups receiving unilateral tDCS in tDCS Sham

INTERVENTIONS:
Device: DLPFC-R (F4) TDCS — direct current brain stimulation- The study was developed through a triple-blind, crossover, randomized, placebo-controlled clinical trial (dummy tDCS). Participants were randomized into three groups receiving unilateral tDCS in DLPFC-L F3 (Block A), combined tDCS in DLPFC-L (F3) and DLPFC-R (F4) simultaneously (Block B) or sham-tDCS (Block C) with equal electrode configuration guaranteed blindness. After the procedures, each participant received the following intervention in the order ABC, BCA or CAB with a period of 1 week between each one. Each block took 3 weeks, organized into: 1) Assessment; 2) Application of stimulation; 3) Reassessment and washout week. Adding 1 more week of final evaluation, the study totaled the period of 10 weeks. During this period, patients were instructed to continue their behavioral/educational treatment and medication routines.
  Arms: DLPFC-L F3 (Block A); tDCS combined in DLPFC-L (F3) and DLPFC-R (F4)
Device: DLPFC-L (F3) and DLPFC-R (F4) TDCS — DLPFC-L (F3) and DLPFC-R (F4) (Bock B)
  Other Names: nibs
  Arms: DLPFC-L F3 (Block A); tDCS combined in DLPFC-L (F3) and DLPFC-R (F4)
Device: sham-tDCS — sham-tDCS (Block C) with equal electrode configuration guaranteed blindness
  Other Names: NIBS
  Arms: DLPFC-L F3 (Block A); tDCS combined in DLPFC-L (F3) and DLPFC-R (F4)

SUMMARY:
To understand the changes in the resting electroencephalogram (EEG) brain networks of children and adolescents with autistic spectrum disorder (ASD) induced by transcranial direct current stimulation (tDCS), we asked two questions. First: how can tDCS modulate the expression of neural network dynamics? Second: how can tDCS modulate functional connections at specific frequencies? We hypothesized that the tDCS mechanism results in increased cortical frequencies in the areas under the anode, which may reflect an increase in synaptic connectivity, and that this tDCS-related increase changes connection profiles at specific frequencies important for ASD, indicating improvement in symptoms. To verify this improvement, the researchers used the Autism Treatment Evaluation Checklist (ATEC) after an intervention, comparing baseline scores with post-treatment scores.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASD reported by a Neuropediatrician; Age group between 5 and 18 years; Mild and moderate clinical symptoms

Exclusion Criteria:

Patients with severe mental illness; Use of a pacemaker or other metal device on the body; Brain tumor or intracranial infection; Uncooperative parents or caregivers; Epilepsy; structural change in the skull

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
to compare the effectiveness of Neuromodulation techniques - transcranial direct current stimulation (tDCS) - in the treatment of people with Autism Spectrum Disorder | 7 weeks
  EEG and TDCS

SECONDARY OUTCOMES:
Check the effects of tDCS modulations on cognitive responses through Autism Treatment Evaluation Checklist | 7 weeks
  ATEC and EEG

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Suellen Marinho Andrade, João Pessoa, Paraíba
  - Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba

IPD SHARING:
Plan to Share IPD: Undecided